CLINICAL TRIAL: NCT00603577
Title: A Multi-center, Randomized, Double Blind, Placebo Controlled Phase III Study to Assess the Efficacy of Xaliproden in Patients With Oxaliplatin-induced Peripheral Sensory Neuropathy (PSN) Following Adjuvant Chemotherapy for Colon Cancer
Brief Title: Role of Xaliproden on Recovery Rate From Severe Neuropathy in Patients Who Have Completed Adjuvant Chemotherapy With Oxaliplatin Based Regimens
Acronym: XENON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: development of product discontinued
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XALIP_C_02090
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — xaliproden

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Xaliproden (Experimental)
  Interventions: Drug: Xaliproden

INTERVENTIONS:
Drug: Placebo — Xaliproden matching placebo. 1 capsule per day for 6 months or until resolution of PSN (whichever comes first).
  Arms: Placebo
Drug: Xaliproden — 1.0 mg capsule. 1 capsule per day for 6 months or until resolution of PSN (whichever comes first).
  Arms: Xaliproden

SUMMARY:
Primary objective:

To assess the effect of xaliproden hydrochloride (xaliproden) 1 mg per oral daily on the rate of complete resolution of peripheral sensory neuropathy (PSN) at 6 months, following randomization, after the completion of oxaliplatin-based adjuvant chemotherapy for colon cancer.

Secondary objective:

* To assess the effect of xaliproden on patient-reported outcomes using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity scale (FACT/GOG NTX-12 subscale).
* To assess the effect of xaliproden on the rate of at least partial recovery of grade > 2 PSN at 6 months
* To assess the effects of xaliproden on the time to complete recovery from PSN
* To evaluate the safety profile of xaliproden

ELIGIBILITY:
Inclusion Criteria:

* Have completed an oxaliplatin-containing chemotherapy regimen post complete surgical removal of primary colon tumor no later than 6 weeks before randomization;
* Have Grade ≥ 1 PSN, as defined by the NCI-CTCAE version 3.0
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2;
* Blood tests within 14 days prior to randomization: (a) AST (SGOT) and ALT (SGPT) ≤2 x upper limit of normal (ULN); (b) serum creatinine ≤1.5 x ULN; (c)HbA1c ≤7%; (d) neutrophils ≥1.5x10^9/L ; (e) platelets ≥50x10^9/L; (f) Serum D-dimer within normal limits

Exclusion Criteria:

* Pre-existing peripheral neuropathy prior to treatment with oxaliplatin
* Receiving any further anti-cancer treatment
* History of any recent (≤1 year) thrombo-embolic events and current clinical evidence of thrombo-embolism
* Unstable cardiac disease
* History of significant neurological or psychiatric disorders including dementia or seizures,
* Active uncontrolled infection
* Active disseminated intravascular coagulation
* Other serious underlying medical conditions which could impair the ability of the patient to participate in the study;
* Use of antidepressant/antiepileptic medication (for the treatment of PSN), unless commenced before informed consent form signed. The addition of these medications (for the treatment of PSN) once the patient has consented is not allowed
* Concurrent treatment with any other experimental drugs
* Pregnant or breast-feeding women;
* Women of childbearing potential must be protected by effective contraceptive methods of birth control. Post-menopausal women must have been amenorrheic for at least 12 months to be considered as having non-childbearing potential
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. Those conditions should be assessed with the patient before registration in the trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Neurological sensory assessment using the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE, Version 3.0) | inclusion, 3 and 6 months and at the 9 and 12 moth follow-up visits

SECONDARY OUTCOMES:
FACT/GOG NTX-12 subscale | AT inclusion and subsequently monthly until month 12
Hematological and biochemical testing | At inclusion, 3 & 6 months
AE graded with NCI-CTCAE (Version 3.0) and coded using Medical Dictionary for Regulatory Activities (MedDRA, version 9.1) | During the whole study period (including follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Principal Investigator — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Québec, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Kallithea, Greece
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom